CLINICAL TRIAL: NCT06842511
Title: Effects on the Anti-inflammatory and Antioxidant Levels of the Adjunctive Use of Hyaluronic Acid-based Gel in the Surgical Periodontal Treatment of Stage III Periodontitis Patients: A Randomized, Split-mouth Clinical Trial
Brief Title: Effects of the Adjunctive Use of Hyaluronic Acid-based Gel in the Surgical Periodontal Treatment of Periodontitis
Acronym: Periodontit
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Prof.Dr. Figen ÖNGÖZ DEDE, Clinical Professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77158231
Record Dates: First submitted 2025-02-06; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Periodontitis (Stage 3)
MeSH Terms: conditions — Periodontitis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): only open flap debridement
  Interventions: Procedure: open flap debridement
- Test group (Active Comparator): open flap debridement + adjunctive use of 0.8% hyaluronic acid-based gel
  Interventions: Drug: open flap debridement and Hyaluronic Acid-Based Gel application; Procedure: open flap debridement

INTERVENTIONS:
Drug: open flap debridement and Hyaluronic Acid-Based Gel application — Hyaluronic Acid-based gel as an adjunctive chemotherapeutic agent
  Other Names: Test group
  Arms: Test group
Procedure: open flap debridement — periodontal surgery technique
  Other Names: Control group

SUMMARY:
This study aimed to assess the effect of Hyaluronic Acid-based gel as an adjunctive chemotherapeutic agent in surgical periodontal treatment on clinical parameters and cytokine levels (IL-6, IL-8, IL-10, IL-17A, TOS, and TAS) in gingival crevicular fluid (GCF) among periodontitis patients.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effects of adjunctive Hyaluronic Acid-Based Gel (HA) application in the surgical treatment of patients with moderate to severe stage III periodontitis (Grade B or C) on clinical parameters, as well as on IL-6, IL-8, IL-10, IL-17, TAS, and TOS levels in gingival crevicular fluid (GCF) to determine its anti-inflammatory and antioxidant efficacy.

This split-mouth study included 18 patients (mean age 43.44±8.12 years) diagnosed with Stage III Grade B or C periodontitis. Quadrants were randomly assigned to two groups: Group 1 (control: open flap debridement [OFD], n=18) and Group 2 (test: OFD + 0.8% HA gel, n=18). Baseline (T0) assessments included plaque index (PI), gingival index (GI), bleeding on probing index (BPI), probing pocket depth (PPD), clinical attachment level (CAL), and GCF collection. Following non-surgical treatment, patients underwent OFD; HA gel was applied to defect sites in the test group and saline in the control. Clinical parameters and GCF sampling were repeated pre-surgery (TS-1), and at 1 month (TS-2) and 6 months (TS-3) post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Stage III Grade B or C periodotitis
* over 18 years old
* signed the informed consent

Exclusion Criteria:

* pregnancy, or lactation,
* systemic problems that would contraindicate for periodontal surgery,
* prosthetic restorations in the test or control teeth,
* taking medications that affect wound healing (corticosteroids, anticancer agents, etc),
* using nonsteroidal anti-inflammatory drugs, using any antibiotics and anti-inflammatory drugs in the last 6 months,
* alcohol abuse and smoking use

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Plaque Index | Baseline
  to assess plaque accumulation
Plaque Index | Pre-surgery
  to assess plaque accumulation
Plaque Index | post-surgery 1 month
  to assess plaque accumulation
Plaque Index | post-surgery 6 months
  to assess plaque accumulation
Gingival Index | Baseline
  for evaluating gingival inflammation
Gingival Index | Pre-surgery
  for evaluating gingival inflammation
Gingival Index | post-surgery 1 month
  for evaluating gingival inflammation
Gingival Index | post-surgery 6 months
  for evaluating gingival inflammation
Probing pocket depth | Baseline
  for measuring disease severity
Probing pocket depth | pre-surgery
  for measuring disease severity
Probing pocket depth | post-surgery 1 months
  for measuring disease severity
Probing pocket depth | post-surgery 6 months
  for measuring disease severity
clinical attachment level | Baseline
  Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
clinical attachment level | pre-surgery
  Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
clinical attachment level | post-surgery 1 months
  Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
clinical attachment level | post-surgery 6 months
  Clinical attachment level (CAL) is calculated by adding or subtracting probing depth (PD) and gingival recession (GR). The formula is CAL = PD + GR. CAL is measured in millimeters.
Bleeding on Probing | baseline
  to assess disease activity
Bleeding on Probing | pre-surgery
  to assess disease activity
Bleeding on Probing | post-surgery 1 months
  to assess disease activity
Bleeding on Probing | post-surgery 6 months
  to assess disease activity
IL-6 | Baseline
  IL-6 levels in gingival crevicular fluid (GCF)
IL-8 | baseline
  IL-8 levels in gingival crevicular fluid (GCF)
IL-17A | baseline
  IL-17A levels in gingival crevicular fluid (GCF)
IL-10 | baseline
  IL-10 levels in gingival crevicular fluid (GCF)
Total antioxidant status | baseline
  TAS levels in gingival crevicular fluid (GCF)
Total oxidant status | baseline
  TOS levels in gingival crevicular fluid (GCF)
IL-6 | pre-surgery
  IL-6 levels in gingival crevicular fluid (GCF)
IL-8 | pre-surgery
  IL-8 levels in gingival crevicular fluid (GCF)
IL-17A | pre-surgery
  IL-17A levels in gingival crevicular fluid (GCF)
IL-10 | pre-surgery
  IL-10 levels in gingival crevicular fluid (GCF)
Total antioxidant status | pre-surgery
  TAS levels in gingival crevicular fluid (GCF)
Total oxidant status | pre-surgery
  TOS levels in gingival crevicular fluid (GCF)
IL-6 | post-surgery 1 month
  IL-6 levels in gingival crevicular fluid (GCF)
IL-8 | post-surgery 1 month
  IL-8 levels in gingival crevicular fluid (GCF)
IL-17A | post-surgery 1 month
  IL-17A levels in gingival crevicular fluid (GCF)
IL-10 | post-surgery 1 month
  IL-10 levels in gingival crevicular fluid (GCF)
Total antioxidant status | post-surgery 1 month
  TAS levels in gingival crevicular fluid (GCF)
Total oxidant status | post-surgery 1 month
  TOS levels in gingival crevicular fluid (GCF)
IL-6 | post-surgery 6 month
  IL-6 levels in gingival crevicular fluid (GCF)
IL-8 | post-surgery 6 month
  IL-8 levels in gingival crevicular fluid (GCF)
IL-17A | post-surgery 6 month
  IL-17A levels in gingival crevicular fluid (GCF)
IL-10 | post-surgery 6 month
  IL-10 levels in gingival crevicular fluid (GCF)
Total antioxidant status | post-surgery 6 month
  TAS levels in gingival crevicular fluid (GCF)
Total oxidant status | post-surgery 6 month
  TOS levels in gingival crevicular fluid (GCF)

CONTACTS AND LOCATIONS:
Overall Officials: Ordu University, Principal Investigator — Ordu University
Locations (1):
- Ordu University, Ordu, Altınordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No